CLINICAL TRIAL: NCT02696915
Title: Fascia Iliaca Compartment Block in Proximal End Femur Fractures, Does it Make a Difference?
Brief Title: Fascia Iliaca Compartment Block for Proximal-end Femur Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS/811
Record Dates: First submitted 2016-02-22; First posted 2016-03-02 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Proximal Femur Fractures
MeSH Terms: conditions — Proximal Femoral Fractures | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients received ultrasound guided fascia iliaca compartment block using 40 ml of saline 0.9%. Then intrathecal medications will be administered.
  Interventions: Drug: Placebo; Device: Ultrasound guided fascia iliaca compartment block; Drug: Intrathecal medications (bupivacaine (15 mg) in conjunction with fentanyl 20 micrograms)
- Bupivacaine (Active Comparator): Patients received ultrasound guided fascia iliaca compartment block using 40 ml of 0.25% bupivacaine. Then intrathecal medications will be administered.
  Interventions: Drug: Bupivacaine; Device: Ultrasound guided fascia iliaca compartment block; Drug: Intrathecal medications (bupivacaine (15 mg) in conjunction with fentanyl 20 micrograms)

INTERVENTIONS:
Drug: Placebo — Patients received ultrasound guided fascial iliaca compartment blockade using normal saline 0.9%, 40 ml
  Arms: Placebo
Drug: Bupivacaine — Patients received ultrasound guided fascial iliaca compartment blockade using bupivacaine 0.25%, 40 ml
  Arms: Bupivacaine
Device: Ultrasound guided fascia iliaca compartment block — Ultrasound guided fascia iliaca compartment block
Drug: Intrathecal medications (bupivacaine (15 mg) in conjunction with fentanyl 20 micrograms) — Intrathecal hyperbaric bupivacaine (15 mg) in conjunction with fentanyl 20 micrograms

SUMMARY:
Fracture femur is a common injury which is associated with excruciating pain. Positioning for neuraxial blocks is always challenging because even slight overriding of the fracture ends is intensely painful .It can causing major patient distress which accompanied by well-known physiological sequelae such as sympathetic activation causing tachycardia, hypotension, and increased cardiac work that may compromise high-risk cardiac patients.

Fascia iliaca compartment block is highly effective in blocking lateral cutaneous nerve of the thigh and femoral nerve. Fascia iliaca compartment block is not only easy to perform but it is also associated with minimal risk as the local anesthetic is injected at a safe distance from the femoral artery and femoral nerve. It is always safe to perform the fascia iliaca compartment block prior to spinal anesthesia as the patient can respond during administration of the local anesthetic and can prevent intra-neuronal injections

DETAILED DESCRIPTION:
On arrival to the pre-operative holding area half hour before the scheduled surgery. Patient will be connected to basal monitoring devices; pulse oximetry and non- invasive blood pressure. Fascia iliaca compartment block will be performed with the aid of ultrasound device in all cases.The injected local anesthetic solution will be prepared by a staff member who was not involved in the study) according to the randomization. After 20 minutes from the injection the investigators will assessed nerves that had been blocked.

On arrival to the operative theater, under complete aseptic technique spinal anesthesia will be carried out in the sitting position (if there is severe pain at positioning we will use lateral position) at space between L3-4 or L4-5 using a 25-gauge spinal quincke needle. After feeling the desired space, the needle will be advanced (paramedian approach) till free flow of cerebrospinal fluid dropped from the needle then 15 mg hyperbaric bupivacaine+20mic fentanyl will be injected.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist physical status I to III
* Patients scheduled for fixation for proximal end femur fracture

Exclusion Criteria:

* Patients refusal
* Morbid obese patients (BMI>40)
* Bleeding diathesis
* Previous femoral bypass surgery
* Inguinal hernia
* Inflammation/infection over injection site
* Peripheral neuropathy
* Allergy to local anesthetics agents used.
* Severely altered consciousness level
* Psychiatric disorders
* Polytrauma

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pain scores | For 24 hours after performance the blockade
  Pain was assessed using visual analogue score

SECONDARY OUTCOMES:
Heart rate | For 24 hours after performance the blockade
Blood pressure | For 24 hours after performance the blockade
Peripheral oxygen saturation | For 24 hours after performance the blockade
Time to performing spinal anesthesia | For 30 min after placement of patient in the optimum position
  Time from the placement of patient in the optimum position to the intra-thecal injection of bupivacaine
Number of trials of dural puncture | For 30 min after placement of patient in the optimum position
Duration of motor blockade | For 12 hours after performing spinal anesthesia
Duration of sensory blockade | For 12 hours after performing spinal anesthesia
Duration of analgesia | For 24 hours after performing spinal anesthesia
  Time from performing spinal anesthesia to first analgesic request
Cumulative consumption of analgesics | For 24 hours after performing spinal anesthesia
  Total opioid or other analgesics received for the first 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Reem A El Sharkawy, MD, Study Chair — Lecturer of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University Hospitals, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043